CLINICAL TRIAL: NCT03745131
Title: A Cohort Study of Serological Responses to MVA-BN Smallpox Vaccine (Imvamex®) Administered During a Monkeypox Outbreak in the UK
Brief Title: Cohort Study of Healthcare Workers Receiving Imvanex®
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Collaborators: Bavarian Nordic (Industry)
Responsible Party: Sponsor
Other Study IDs: MPX Imvanex Serology; 18/LO/1957 (Other: London-West London & GTAC Research Ethics Committee); 255382 (Other: Integrated Research Application System)
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2018-11

CONDITIONS: Monkeypox
Keywords: Immunisation; Modified Vaccinia Ankara; Imvanex; Imvamune; Vaccine
MeSH Terms: conditions — Mpox, Monkeypox | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-exposure prophylaxis recipients: 40 healthcare workers who provide specialist medical care to patients with monkeypox and who received vaccine as pre-exposure prophylaxis.
  Interventions: Other: Blood draw
- Post-exposure prophylaxis recipients: 40 healthcare workers who received vaccine as post-exposure prophylaxis following monkeypox-exposure risk assessments.
  Interventions: Other: Blood draw
- Control Group 1: 20 healthcare workers who provided specialist medical care to patients with monkeypox but declined the offer of vaccine as pre-exposure prophylaxis.
  Interventions: Other: Blood draw
- Control Group 2: Healthcare workers not involved in the care of, and have not had known exposure to, patients with monkeypox and, therefore, were not offered vaccine.
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood draw to obtain serum to determine anti-orthopox antibody titres.

SUMMARY:
During an outbreak of monkeypox in the UK in 2018, a third generation smallpox vaccine, Imvanex, was used for the first time to immunise healthcare workers who had been, or were expected to be, in contact with cases of monkeypox. This study will examine the antibody responses in these healthcare workers compared to control groups, to provide evidence that the vaccine can produce a response consistent with protection when used in this context.

DETAILED DESCRIPTION:
This study intends to describe antibody responses to a third generation smallpox vaccine, Imvanex® (MVA-BN, Bavarian Nordic GmBH; also known as Imvamune®), in cohorts of individuals who received the vaccine for pre-exposure or post-exposure prophylaxis against monkeypox during a monkeypox outbreak in the UK. In addition to quantifying anti-vaccinia virus antibody responses to vaccine, the study intends to demonstrate that vaccine-induced antibodies neutralise the specific monkeypox viruses involved in the UK outbreak, and also reference monkeypox viruses. The use of Imvanex® during the UK outbreak represents the first ever use of Imvanex® as a public health intervention for a monkeypox outbreak, and this study will provide an opportunity to quantify and characterise antibody responses to Imvanex® administered in a non-trial setting.

ELIGIBILITY:
Inclusion criteria for pre-exposure prophylaxis cases:

* A High Consequence Infectious Disease (HCID) Centre healthcare worker involved in the care of a confirmed monkeypox case
* AND the individual has received Imvanex® during the outbreak period
* AND no known unprotected exposure to a monkeypox case (i.e. pre-exposure indication for vaccination)

Inclusion criteria for post-exposure prophylaxis cases:

* A healthcare worker
* AND the individual has received Imvanex® during the outbreak period
* AND unprotected exposure to a monkeypox case is believed to have occurred (i.e. post-exposure indication for vaccination)

Inclusion criteria for control group 1 (unvaccinated HCID staff caring for confirmed cases):

* A High Consequence Infectious Disease (HCID) Unit healthcare worker involved in the care of a confirmed monkeypox case
* AND the individual has NOT received Imvanex® during the outbreak period
* AND no known unprotected exposure to a monkeypox case

Inclusion criteria for control group 2 (general healthcare workers):

* A healthcare worker NOT involved in the care of a confirmed monkeypox case
* AND the individual has NOT received Imvanex® during the outbreak period
* AND no known unprotected exposure to a monkeypox case

Exclusion criteria for all participants:

* Refusal by participant
* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers at NHS Airborne HCID Centres, and healthcare workers at other NHS hospitals that cared for monkeypox cases before they were transferred to HCID Centres.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Antibody responses to first dose of Imvanex® | 28-56 days following immunisation
  The proportion of participants with anti-orthopox antibodies when measured at a single time point between days 28 and 56 following first dose of Imvanex®.
Antibody titres following first dose of Imvanex® | 28-56 days following immunisation
  Geometric mean titres (GMTs) of anti-orthopox antibodies when measured at a single time point between days 28 and 56 following first dose of Imvanex®.

SECONDARY OUTCOMES:
Antibody responses to second dose of Imvanex® | 28-56 days following immunisation
  The proportion of participants who have anti-orthopox antibodies when measured at day 14 following the second dose of Imvanex®, if a subset of individuals receive a second dose of Imvanex® during the lifetime of the study.
Antibody titres following second dose of Imvanex® | 28-56 days following immunisation
  The geometric mean titres (GMTs) of anti-orthopox antibodies when measured at day 14 following the second dose of Imvanex®, if a subset of individuals receive a second dose of Imvanex®.
Neutralising antibody responses to first dose of Imvanex® | 28-56 days following immunisation
  The proportion of participants who have demonstrable neutralising antibodies against the specific monkeypox viruses involved in the UK outbreak, in addition to reference monkeypox viruses.
Adverse events reported following vaccination with Imvanex® | 28-56 days following immunisation
  Adverse events and serious adverse events by reported frequencies (reported retrospectively).

CONTACTS AND LOCATIONS:
Overall Officials: William Jake Dunning, MRCP PhD, Study Director — Public Health England; Meera Chand, FRCPath, Study Director — Public Health England; Sema Mandal, MRCP FFPH, Principal Investigator — Public Health England; Nicholas Andrews, PhD, Principal Investigator — Public Health England; Timothy Brooks, FRCPath, Principal Investigator — Public Health England; Michael Beadsworth, MD MRCP, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust; Michael Jacobs, FRCP PhD, Principal Investigator — Royal Free London NHS Foundation Trust; Matthias Schmid, MD FRCP, Principal Investigator — Newcastle Hospitals NHS Foundation Trust; Christopher Meadows, FRCP FRCA, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Peter Flegg, MD FRCP, Principal Investigator — Blackpool Teaching Hospitals NHS Foundation Trust; Heinz Weidenthaler, Principal Investigator — Bavarian Nordic
Locations (5):
- United Kingdom (5):
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, Lancashire
  - Royal Liverpool and Broadgreen University Hospitals NHS Trust, Liverpool, Merseyside
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - Royal Free London NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vaughan A, Aarons E, Astbury J, Balasegaram S, Beadsworth M, Beck CR, Chand M, O'Connor C, Dunning J, Ghebrehewet S, Harper N, Howlett-Shipley R, Ihekweazu C, Jacobs M, Kaindama L, Katwa P, Khoo S, Lamb L, Mawdsley S, Morgan D, Palmer R, Phin N, Russell K, Said B, Simpson A, Vivancos R, Wade M, Walsh A, Wilburn J. Two cases of monkeypox imported to the United Kingdom, September 2018. Euro Surveill. 2018 Sep;23(38):1800509. doi: 10.2807/1560-7917.ES.2018.23.38.1800509. PMID 30255836
- [Derived] Hatmal MM, Al-Hatamleh MAI, Olaimat AN, Ahmad S, Hasan H, Ahmad Suhaimi NA, Albakri KA, Abedalbaset Alzyoud A, Kadir R, Mohamud R. Comprehensive literature review of monkeypox. Emerg Microbes Infect. 2022 Dec;11(1):2600-2631. doi: 10.1080/22221751.2022.2132882. PMID 36263798
- See also: Public Health England News Story: Monkeypox case in England (update) — https://www.gov.uk/government/news/monkeypox-case-in-england